CLINICAL TRIAL: NCT05828966
Title: HUMAN CHORIONIC GONADOTROPIN (HcG) VS MAGNESIUM SULPHATE (MgSo4) AS A TOCOLYTIC AGENT- A RANDOMIZED CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Hafiza Faiza Mushtaq, Resident in Gynecology and Obstetrics, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Chorionic Gonadotropin; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HUMAN CHORIONIC GONADOTROPIN (HCG) Group (Active Comparator): H.C.G. will be given in Group A and in a dose of 5000units intramuscular injection followed by a drip of 10,000 units in 500ml of dextrose 5%, at the rate of 20 drops per minute. Half hourly assessment of uterine contractions, maternal vital signs, fetal heart rate monitoring will be done.
  Interventions: Drug: human chorionic gonadotropin (hCG)
- Magnesium Sulphate(MgSO4) Group (Active Comparator): 4gm of MgSO4 will be given in Group B as intravenously as continuous dose followed by 2gm/hr till uterine quiescence is achieved.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: human chorionic gonadotropin (hCG) — H.C.G. will be given in Group A and in a dose of 5000units intramuscular injection followed by a drip of 10,000 units in 500ml of dextrose 5%, at the rate of 20 drops per minute.
  Arms: HUMAN CHORIONIC GONADOTROPIN (HCG) Group
Drug: Magnesium sulfate — 4gm of MgSO4 will be given in Group B as intravenously as continuous dose followed by 2gm/hr till uterine quiescence is achieved.
  Arms: Magnesium Sulphate(MgSO4) Group

SUMMARY:
Preterm labor is defined as regular contractions of the uterus resulting in changes in the cervix (effacement and dilatation) that start before 37 weeks of pregnancy. (1) Although preterm labor constitutes only 10% of total labors, yet 70% of infant's mortality is related to prematurity. It is therefore one of the international indices in assessment of health condition worldwide. Human Chorionic Gonadotropin (H.C.G.) is a heterodimeric glycoprotein produced primarily in the placenta and has multiple endocrines, paracrine and immunoregulatory actions. (3) The importance of H.C.G. in maintenance of early pregnancy has been widely accepted, reports have highlighted a potential role of H.C.G. in maintaining uterine quiescence in the third trimester. H.C.G. exerts a potent concentration dependent inhibitory effect on human myometrial contractions. (4) Recent data suggests that H.C.G. might have a role as an endogenous tocolytic agent in normal pregnancy. A significant decrease in serum H.C.G. level was found 2-3 weeks before the spontaneous onset of labour. This might contribute to increasing the contractility in the uterine muscle and gradually initiating the onset of labour. (5)

DETAILED DESCRIPTION:
Preterm labor is defined as regular contractions of the uterus resulting in changes in the cervix (effacement and dilatation) that start before 37 weeks of pregnancy. (1) Although preterm labor constitutes only 10% of total labors, yet 70% of infant's mortality is related to prematurity. It is therefore one of the international indices in assessment of health condition worldwide. Factors that increase the risk of preterm birth include history of previous preterm birth, short cervix, short time between pregnancies, teenage pregnancy, history of certain types of surgery on the uterus or cervix, certain pregnancy complications, such as multiple pregnancy and vaginal bleeding and lifestyle factors such as low pre-pregnancy weight, smoking during pregnancy, and substance abuse during pregnancy.

Preterm labor can be diagnosed clinically only when changes in the cervix are found after pelvic examination along with contractions also may be monitored. A transvaginal ultrasound exam may be done to measure the length of your cervix. Tocolytics are drugs used to delay delivery for a short time (up to 48 hours). They may allow time for corticosteroids or magnesium sulfate to be given or for you to be transferred to a hospital that offers specialized care for preterm infants. (1,2) Tocolytic agents are β- HCG, MgSO4, nifedipine, β-agonists(salbutamol) and atosiban. Use of salbutamol is of limited use because of many cardiovascular complications i.e., ventricular arrythmia, hypertension and hyperglycemia while atosiban is expensive and not available in Pakistan.

Human Chorionic Gonadotropin (H.C.G.) is a heterodimeric glycoprotein produced primarily in the placenta and has multiple endocrines, paracrine and immunoregulatory actions. (3) The importance of H.C.G. in maintenance of early pregnancy has been widely accepted, reports have highlighted a potential role of H.C.G. in maintaining uterine quiescence in the third trimester. H.C.G. exerts a potent concentration dependent inhibitory effect on human myometrial contractions. (4) Recent data suggests that H.C.G. might have a role as an endogenous tocolytic agent in normal pregnancy. A significant decrease in serum H.C.G. level was found 2-3 weeks before the spontaneous onset of labour. This might contribute to increasing the contractility in the uterine muscle and gradually initiating the onset of labour. (5) Following I.M. injection, peak concentration of H.C.G. occurs about 6 hrs after a dose. It is distributed primarily to gonads. Blood concentration declines in a biphasic manner, with a half-life between about 6 and 11 hrs and 23 to 38 hrs respectively. About 10 to 12% of an IM dose is excreted in urine within 24 hours. (6)

ELIGIBILITY:
Inclusion Criteria:

1. 4 uterine contractions per 20 min or 8 contractions per hour
2. single live fetus
3. Pregnancy less than 37 weeks
4. Intact Membranes,
5. Dilatation less than 3cm and effacement less than 80%.

Exclusion Criteria:

1. Cervical Dilatation more than 4 cm
2. Abnormal vaginal bleeding
3. Premature Rupture of membranes
4. Cardiopulmonary compromised
5. Fetal and Uterine anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant females
Enrollment: 70 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Tocolysis | 48 hours
  Tocolysis will be considered successful when contractions ceased and delivery will be delayed by 48 hrs giving time to the administered corticosteroids to accelerate fetal lung maturation

CONTACTS AND LOCATIONS:
Locations (1):
- Mother and Child Care Hospital, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
I have not decided yet .